CLINICAL TRIAL: NCT03534700
Title: Excision and Reconstruction of the Natal Cleft With a Parasacral Perforator Flap Versus Open Excision With Secondary Healing, in the Management of Sacrococcygeal Pilonidal Disease. A Randomized Controlled Study.
Brief Title: Excision and Reconstruction of the Natal Cleft With a Parasacral Perforator Flap Versus Open Excision With Secondary Healing, in the Management of Sacrococcygeal Pilonidal Disease.
Acronym: PILOPERFO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decision of the PI
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/16/8255
Record Dates: First submitted 2017-11-24; First posted 2018-05-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Pilonidal Disease
Keywords: sacrococcygeal pilonidal disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open excision (Active Comparator): open excision and healing by secondary intention, marsupialization, excision and primary closure (midline or off-midline), excision and repair by flap.
  Interventions: Procedure: open excision
- parasacral flap reconstruction (Experimental): The parasacral perforator flap has been described. It appears to be a good alternative, offering all the benefits of the reconstruction of the natal cleft in terms of lower rate of recurrence and lower time for complete wound healing. It also gives a better aesthetic result.
  Interventions: Procedure: parasacral flap reconstruction

INTERVENTIONS:
Procedure: parasacral flap reconstruction — parasacral flap reconstruction
  Arms: parasacral flap reconstruction
Procedure: open excision — open excision and healing by secondary intention, marsupialization, excision and primary closure (midline or off-midline), excision and repair by flap.
  Arms: Open excision

SUMMARY:
Chronic sacrococcygeal pilonidal disease is a common acquired condition associated with hirsutism that predominantly affects young male patients. Morbidity from this disease results in pain, embarrassment and loss of normal activities, causing absenteeism from work and school.

Various surgical procedures have been described for the treatment of both primary and recurrent pilonidal disease counting: open excision and healing by secondary intention, marsupialization, excision and primary closure (midline or off-midline), excision and repair by flap.

No single method has been accepted as the "gold standard", and none of them cancels the risk of recurrence.

The optimal therapy for pilonidal sinus disease should be simple, with good aesthetic outcomes and a low recurrence rate. It must allow the return to normal activities quickly.

The parasacral perforator flap seems to answer these entire requirements. No study compares this flap repair with the most common procedure, which is the open excision with secondary healing. The aim of this study is to assess the efficacy and the security of the reconstruction of the natal cleft with the perforator parasacral flap versus open excision with secondary healing in the treatment of sacrococcygeal pilonidal sinus.

DETAILED DESCRIPTION:
Many studies seem to attest the superiority of excision and reconstruction of the natal cleft with a flap rather than the open excision with secondary healing. Jamal et al. found a significantly lower recurrence rate with a rhomboid excision and reconstruction with a Limberg flap versus open excision and secondary healing (p=0.005) in a prospective controlled randomized trial including 49 patients. Keshuari et al. obtained the same significant results in their prospective controlled randomized study including 321 patients, with a rate of 1.2% of recurrence in the Karidakis flap repair cluster versus 7.5% in the excision with healing by secondary intention cluster. The time for complete wound healing was also significantly amended .

The reconstruction of the natal cleft with a Karydakis or Limberg flap seemed to be superior in terms of recurrence compared to open excision. But those flaps led to a significant and discernable scar.

The parasacral perforator flap has been described by Garrido et al. in 2002. It appears to be a good alternative, offering all the benefits of the reconstruction of the natal cleft in terms of lower rate of recurrence and lower time for complete wound healing. It also gives a better aesthetic result.

In this trial, patients will be operated under general anesthesia. A Methylene blue injection will identify the limits of the pilonidal sinus. An excision of the whole width of the relevant area will be performed, with depth reaching the presacral fascia. In the A group, a parasacral perforator flap repair of the natal clef will be done, and in the B group healing by secondary intention by dressing will be performed. Patients will be followed in consultation at 15 days, 3 months, 6 months, 1 year and 2 years.

During these visits, a potential clinical recurrence will be detected, the time to be completely healing will be evaluated, the period of loss of normal activities will be noted, the quality of life will be assessed by a standardized generic measure (EQ-5D-5L) and by a specific score (DLQI), and post-operative complications will be collected.

The aim of this study is to assess the efficacy and the security of the reconstruction of the natal cleft with the perforator parasacral flap versus open excision with secondary healing in the treatment of sacrococcygeal pilonidal sinus.

A medico-economic analysis evaluating the incremental cost-effectiveness and cost-utility ratio will be also done at 2 years. Additionally, an evaluation of the production costs of the new strategy (i.e. parasacral perforator flap) will be performed from the specific perspective of hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary or recurrent sacrococcygeal pilonidal sinus disease,
* Minimum delay of 1 month after an infection of the pilonidal areas,

Exclusion Criteria:

* Florid abcess in the pilonidal sinus,
* Impossibility of general anesthesia, allergy to methylene blue, anticoagulant therapy,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
recurrence | 2 years
  the rate of recurrence during a follow up of 2 years.

SECONDARY OUTCOMES:
cost-effectiveness | 2 years
  Incremental cost-effectiveness evaluation of comparative perforation flap surgery to the reference strategy in patients with pilonidal sinus cysts : the number of recurrences at 24 month
cost-utility | 2 years
  Incremental cost-utility ratios

CONTACTS AND LOCATIONS:
Overall Officials: Benoit CHAPUT, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital, Montpellier
  - University hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No